CLINICAL TRIAL: NCT07402603
Title: Enhancing Patient Care: Sleep and Ventilation Database
Brief Title: Sleep-disordered Breathing Database
Status: Not yet recruiting | Type: Observational
Sponsor: Royal Free Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 25-WS-0157
Record Dates: First submitted 2026-01-13; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Obstructive Sleep Apnoea (OSA); Hypoventilation Syndrome
Keywords: database; observational
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sleep disordered breathing: Patients who are referred for a sleep study to investigate sleep disordered breathing

SUMMARY:
The goal of this study is to collect clinical data on patients who have had a sleep study and are given a diagnosis of a sleep related breathing disorder such as obstructive sleep apnoea. Collecting this data in an organised way will mean that the investigators can monitor patients and their health outcomes.

DETAILED DESCRIPTION:
This is a prospective database collecting: symptom, physiological, comorbidity and treatment response data

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Referred to Royal Free London NHS Foundation Trust Sleep and Ventilation Service
* Agreed to undertake a sleep study

Exclusion Criteria:

* Inability to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The patient population will be those patients under the sleep and ventilation service who have undertaken a sleep study and started on treatment for their sleep disordered breathing
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2031-01-14 (Estimated); Study Completion 2036-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients consenting to participation in a database | 5 years
  From the whole cohort referred for a sleep study, the number of participants (percentage of the whole cohort) who sign a consent form and have data recorded will be calculated

SECONDARY OUTCOMES:
Changes in symptoms and disease related variables | 5 years initially, further ethical approval will be sought at 5 years to extend the database further
  Changes in symptom based scores - Epworth sleepiness score between baseline and follow up Changes in disease parametrics including: AHI (apnoea/hypopnoea index), blood gas measurements (PO2, PCO2, pH, HCO3), lung function between baseline and follow up Additional variables may be added over the duration of the database

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Free London NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Other researchers may apply for access to the database, provided they demonstrate a valid scientific and public benefit and meet all governance requirements.